CLINICAL TRIAL: NCT03786393
Title: Investigation of Estrogen Receptor 1 Gene Polymorphism Frequency in Patients With Fibromyalgia Syndrome
Brief Title: Estrogen Receptor 1 Gene Polymorphism Frequency in Fibromyalgia Syndrome
Status: Completed | Type: Observational
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Ercan KAYDOK, Assistant of Proffessor M.D. Ercan Kaydok, Nigde Omer Halisdemir University
Other Study IDs: Nigde O.H.U.
Record Dates: First submitted 2018-12-20; First posted 2018-12-26 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-01

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Migraine; estrogen receptor alpha; polymorphism
MeSH Terms: conditions — Fibromyalgia; Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Estrogen receptor alpha polymorphism
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fibromyalgia: 100 participants diagnosed with fibromyalgia according to ACR 1990 criteria.
  Interventions: Diagnostic Test: ACR 1990 fibromyalgia critters
- Control
  Interventions: Diagnostic Test: ACR 1990 fibromyalgia critters

INTERVENTIONS:
Diagnostic Test: ACR 1990 fibromyalgia critters — ACR 1990 fibromyalgia critters

SUMMARY:
Fibromyalgia Syndrome (FMS) is a chronic musculoskeletal disorder accompanied by diffuse body pain, increased fatigue and tenderness in specific anatomical regions, and sleep disturbance. The higher prevalence of FMS in women and the observation of it from young adulthood suggest the effect of sex hormones on the pathophysiology of this condition. Steroid hormones, especially estrogen, have effects on both the peripheral and central nervous system receptors (estrogen receptor-a [ERa] and estrogen receptor-b [ERb]), on the inflammatory process, and on central pain delivery. However, the mechanism of action of these hormonal effects is still unknown and is a matter of debate.

The fact that fibromyalgia syndrome and migraine are more common in women of reproductive age and their incidence is higher than other populations suggests that these two diseases may have a common genetic basis. Previous studies have shown that ESR-1 594G> A (rs2228480), ESR-1 325C> G (rs2295190) polymorphisms significantly increase the risk of migraine occurrence. However, there are no studies investigating these polymorphisms in FMS. In this study, it was aimed to investigate whether there is a relationship between ESR-1 594G> A (rs2228480) and ESR-1 325C> G (rs2295190) polymorphisms and fibromyalgia disease.

DETAILED DESCRIPTION:
Objective: The fact that fibromyalgia and migraine are more common in women of reproductive age and their incidence are higher than other populations suggests that these three diseases may have a common genetic basis. Therefore, we aimed to investigate whether there is a relationship between ESR-1 594G> A (rs2228480), ESR-1 325C> G (rs2295190) polymorphisms and fibromyalgia disease.

Introduction: Fibromyalgia syndrome (FMS), diffuse body pain, chronic musculoskeletal disease with increased fatigue and tenderness and sleep disorder in specific anatomical regions . The FMS diagnosis is based on American College of Rheumatology(ACR) 1990 classification criteria. FM frequently affects women between 30 and 50 years of age and its prevalence is between 1% and 4% of the whole population, 0-4% in men and 2.5-10.5% in women. Researchers have found that the strong familial tendency in FM has a risk of developing FM in first-degree relatives of patients with FM, 8 times more than in the general population. Family members of FM patients are more susceptible to pain and are more likely to develop conditions such as irritable bowel syndrome (IBS), temporomandibular disorder (TMD), headache-migraine, restless leg syndrome, and other regional pain syndromes . Several studies have been conducted to demonstrate specific genetic polymorphism in FM. To date, polymorphisms in the serotonin receptor, serotonin transporter, dopamine D4 receptor and catechol-O-methyltransferase genes have been found to be high . All these identified polymorphisms are responsible for the metabolism and transport of monoamines; These are compounds that play a critical role in the human stress response.

The more frequent occurrence of FMS in women is observed in young adults, indicating the effect of sex hormones on the pathophysiology of this condition. However, the mechanism of action of these hormonal effects is still unknown and is a matter of debate. Steroid hormones, in particular estrogen, affect both peripheral and central nervous system (CNS) receptors (Estrogen Receptor-1; estrogen receptor-a [Era] and Estrogen Receptor-2;estrogen receptor-b [ERb]), the inflammatory process and the transmission of central pain. For example, estrogen may directly affect monocytes and macrophages to regulate the production of cytokines (eg, Interleukin-1 [IL-1], IL-6 and tumor necrosis factor-a [TNF-a]).

Migraine is a neurological disorder characterized by episodes of hemicranial pain characterized by attacks. one-year prevalence of migraine in the general population in Turkey 16.4%, while the proportion of patients with FM were significantly lower (9). The incidence of headache increased in patients with fibromyalgia syndrome. Migraine and non-migraine headaches have been reported in patients with FM between 28% and 58% . Similarly, in a study conducted on 33 FM patients, the current migraine was present at 45% and the lifetime migraine history was 55% . The prevalence of migraine has been reported to be approximately 2-fold (reproductive period) and the severity of migraine attacks in women compared to men . Studies investigating the relationship between sex hormone levels and polymorphisms due to more frequent reproductive states have shown that they are associated with estrogen receptor-alpha (ERa 594G> A (rs2228480), ERa 325C> G (rs2295190) polymorphisms.

Methods: Establishment of study groups: 100 patients diagnosed as Fibromyalgia syndrome according to the criteria of ACR 1990, 18-65 years old, and having similar sociodemographic characteristics. 100 control patients will be taken. As the inclusion criteria for the patients; Being between 18 and 60 years of age, taking the diagnosis of primary FMS according to ACR 1990 diagnostic criteria, accepting to participate in the study, lack of any sex hormone disease. The control group will be composed of volunteers with similar age and gender characteristics. The volunteers taken into the control group will have no sex hormone. The participants will be informed about the subject before being taken into the study and the necessary permits will be taken.

Semi-structured sociodemographic information form prepared by us will be used in accordance with the clinical experience and the information obtained from the scanned sources and the aims of the study (ANNEX-1) Age, gender, education level, marital status, BMI, family history of fibromyalgia diseases and accompanying symptoms. Accompanied by the symptoms; TMD symptoms such as migraine type headache, jaw pain and locking, sleep disorder, dry mouth, dry eyes, irritable bowel symptoms, restless leg symptoms, soft tissue swelling, fatigue, depressive symptoms or depression history will be questioned. Patients with headache will be evaluated by a neurologist in terms of the diagnosis of migraine. Pain evaluation of the cases will be done by Visual Analog Scale (VAS). A 10 cm ruler will be used for this. Patients will be evaluated once and the appropriate amount of blood samples will be collected from the patients after the evaluation.

Collection of Blood Samples: 5 mL blood samples from the control and patient groups will be taken into sterile, citrate tubes. The blood in the tubes will be stored at -80 ° C until isolation of the DNA.

Isolation of Genomic DNA: Genomic DNA will be isolated from the blood using a DNA isolation kit. DNA purity will be determined by spectrophotometric method.

Genotyping: Genotyping of ESR-1 325 C> G and 594 G> A polymorphisms in the study group will be performed by using single nucleotide polymorphism analysis kit and sequence-specific double-dye hydrolysis probes and allelic segregation analysis in real-time polimerase chain reaction (RT-PCR) using primers. Genotyping of each patient and control will be repeated 3 times to ensure the reliability of the analysis results.

Statistical methods: The number of individuals to be included in the study was determined by Statistical Power Analysis. In this study, when α = 0.05, β = 0.10, 1- β = 0.90, it was decided to take 100 individuals to each patient and control groups, and the strength of the test was found to be p = 0.9072. All data obtained from the study will be evaluated with SPSS 18 program. The χ2 test and Student-t and Mann-Whitney tests will be used to evaluate the suitability of nominal and continuous variables.

ELIGIBILITY:
---Inclusion Criteria: As the inclusion criteria for the Fibromyalgia group ;

* Being between 18 and 60 years of age,
* Taking the diagnosis of primary FMS according to ACR 1990 diagnostic criteria,
* Accepting to participate in the study

As the inclusion criteria for the Control group;

* Being between 18 and 60 years of age,
* Accepting to participate in the study
* No diagnosis of fibromyalgia.

  ---Exclusion Criteria:
* Having any sex hormone disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Fibromyalgia: 100 person, Control: 100 person.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
polymorphism frequency | 9 month
  The frequency of estrogen receptor alpha polymorphism in fibromyalgia and control group

CONTACTS AND LOCATIONS:
Locations (1):
- BOR Physical medicine and rehabilitaton hospital, Niğde, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bradley LA, Alarcon GS. Fibromyalgia. In: Kopman WJ (ed). Arthritis and Allied Conditions. Philedelphia. Lippincott & Williams & Wilkins, 2001, 1811-44.
- [Background] Wolfe F, Smythe HA, Yunus MB, Bennett RM, Bombardier C, Goldenberg DL, Tugwell P, Campbell SM, Abeles M, Clark P, et al. The American College of Rheumatology 1990 Criteria for the Classification of Fibromyalgia. Report of the Multicenter Criteria Committee. Arthritis Rheum. 1990 Feb;33(2):160-72. doi: 10.1002/art.1780330203. PMID 2306288
- [Background] Ertas M, Baykan B, Orhan EK, Zarifoglu M, Karli N, Saip S, Onal AE, Siva A. One-year prevalence and the impact of migraine and tension-type headache in Turkey: a nationwide home-based study in adults. J Headache Pain. 2012 Mar;13(2):147-57. doi: 10.1007/s10194-011-0414-5. Epub 2012 Jan 14. PMID 22246025
- [Background] Lipton RB, Stewart WF, Diamond S, Diamond ML, Reed M. Prevalence and burden of migraine in the United States: data from the American Migraine Study II. Headache. 2001 Jul-Aug;41(7):646-57. doi: 10.1046/j.1526-4610.2001.041007646.x. PMID 11554952
- [Background] Schurks M, Rist PM, Kurth T. Sex hormone receptor gene polymorphisms and migraine: a systematic review and meta-analysis. Cephalalgia. 2010 Nov;30(11):1306-28. doi: 10.1177/0333102410364155. Epub 2010 May 4. PMID 20959426
- [Background] Headache Classification Subcommittee of the International Headache Society. The International Classification of Headache Disorders: 2nd edition. Cephalalgia. 2004;24 Suppl 1:9-160. doi: 10.1111/j.1468-2982.2003.00824.x. No abstract available. PMID 14979299
- [Background] Hudson JI, Goldenberg DL, Pope HG Jr, Keck PE Jr, Schlesinger L. Comorbidity of fibromyalgia with medical and psychiatric disorders. Am J Med. 1992 Apr;92(4):363-7. doi: 10.1016/0002-9343(92)90265-d. PMID 1558082
- [Background] Clark S, Campbell SM, Forehand ME, Tindall EA, Bennett RM. Clinical characteristics of fibrositis. II. A "blinded," controlled study using standard psychological tests. Arthritis Rheum. 1985 Feb;28(2):132-7. doi: 10.1002/art.1780280204. PMID 3882093